CLINICAL TRIAL: NCT03589482
Title: Assessing Lung Inhomogeneity During Ventilation for Acute Hypoxemic Respiratory Failure
Acronym: ALIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-6091; 17-6226 (Other: UHN CAPCR Related ID)
Record Dates: First submitted 2018-04-06; First posted 2018-07-18 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2020-08

CONDITIONS: Acute Respiratory Distress Syndrome; Mechanical Ventilation Pressure High; Hypoxemic Respiratory Failure
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EIT algorithm (Experimental): Patients randomized to this arm will be ventilated at the PEEP level selected by the EIT algorithm, which selects a PEEP at which both collapse and hyperdistention are minimized.
  Interventions: Device: Electrical Impedance Tomography
- ExPRESS algorithm (Active Comparator): Patients randomized to this arm will be ventilated at the PEEP level selected by the ExPRESS algorithm, which is a method that targets a tidal volume of 6 ml/kg predicted body weight and then titrates PEEP until plateau airway pressure reaches 28 cm H2O.
  Interventions: Other: ExPRESS-derived PEEP level

INTERVENTIONS:
Device: Electrical Impedance Tomography — Electrical impedance tomography (EIT) is a new technique that enables real-time visualization of the distribution of ventilation at the bedside. This technique allows clinicians and investigators to immediately determine how applying higher or lower PEEP levels affect stress and strain in the lung. The investigators propose to apply this new technique to test a strategy for finding the optimal level of PEEP that prevents lung injury and improves outcomes in critically ill patients.
  Arms: EIT algorithm
Other: ExPRESS-derived PEEP level — The ExPRESS algorithm is a traditional approach to selecting PEEP based on respiratory mechanics.
  Arms: ExPRESS algorithm

SUMMARY:
Mechanical ventilation can cause damage by overstretching the lungs, especially when the lungs are collapsed or edematous. Raising ventilator pressures can reduce lung collapse and this can prevent overstretching from mechanical ventilation. It remains uncertain how much pressure (PEEP - positive end-expiratory pressure) should be used on the ventilator and how to identify patients who will benefit from higher ventilator pressures vs. lower ventilator pressures. The investigators are using a unique new imaging technology, electrical impedance tomography (EIT), to study this problem and to determine the safest and most effective ventilator pressure level. The results of this study will inform future trials of higher vs. lower PEEP strategies in mechanically ventilated patients.

DETAILED DESCRIPTION:
Patients participating in this physiological cross-over randomized trial will undergo a series of PEEP maneuvers designed to assess lung recruitability, PEEP responsiveness, and optimal PEEP. EIT imaging and esophageal manometry will be employed throughout the protocol to quantify the effect of PEEP on lung function. Patients will be randomized to be ventilated at PEEP levels supplied by the ExPRESS strategy or by the EIT hyperdistention/collapse algorithm. The biological response will be assessed by measuring serum cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Acute (≤7 days) hypoxemia with PaO2:FiO2 ratio less than or equal to 200 mm Hg
* Oral endotracheal intubation and mechanical ventilation
* Bilateral airspace opacities on chest radiograph or CT

Exclusion Criteria:

* Contraindication to EIT electrode placement (burns, chest wall bandaging limiting electrode placement)
* Contraindication to esophageal catheter placement (recent upper GI surgery, actively bleeding esophageal varices)
* Respiratory failure predominantly due to cardiogenic cause or fluid overload
* Ongoing hemodynamic instability (requiring 2 vasopressor agents by continuous infusion AND rising vasopressor infusion rate requirements in the previous 8 hours)
* Ongoing ventilatory instability (P/F < 70 mm Hg, pH < 7.2; ventilator driving pressures, PEEP, or FiO2 increasing by more than 25% in previous 30 minutes)
* Intracranial hypertension (suspected or diagnosed by medical team)
* Known or suspected pneumothorax recognized within previous 72 hours
* Bronchopleural fistula
* Bridge to lung transplant
* Recent lung transplantation (within previous 6 weeks)
* Attending physician deems the transient application of high airway pressures (>40 cm H2O) to be unsafe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Intratidal ventilation heterogeneity | Assessed after completion of 3 hours on randomized strategy (EIT vs ExPRESS)
  A measure of variation in the distribution of ventilation throughout the lung as detected by electrical impedance tomography

SECONDARY OUTCOMES:
Difference in the optimal PEEP levels identified by several different PEEP titration strategies | Assessed immediately after completion of decremental PEEP titration procedure
  Compare the relative degree of agreement or disparity between PEEP levels recommended by different PEEP titration strategies
Change in ratio of partial pressure of oxygen (PaO2) to inspired fraction of oxygen (FiO2) ratio following a standardized increased in PEEP | Assessed 10 minutes after step PEEP increase from 6-8 to 16-18 cm H2O
  Measurement of changes in oxygenation by PaO2/FiO2 ratio due to PEEP
Respiratory mechanics (transpulmonary driving pressure) | Assessed after completing 3 hours on the randomized PEEP strategy (EIT vs ExPRESS)
  The swing in transpulmonary pressure during inspiration, a measure of dynamic lung stress

CONTACTS AND LOCATIONS:
Overall Officials: Ewan Goligher, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santa Cruz R, Villarejo F, Irrazabal C, Ciapponi A. High versus low positive end-expiratory pressure (PEEP) levels for mechanically ventilated adult patients with acute lung injury and acute respiratory distress syndrome. Cochrane Database Syst Rev. 2021 Mar 30;3(3):CD009098. doi: 10.1002/14651858.CD009098.pub3. PMID 33784416